CLINICAL TRIAL: NCT01328145
Title: Acetylic Salicylic Acid for the Treatment of Chronic Obstructive Pulmonary Disease (COPD). A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Acetylic Salicylic Acid for the Treatment of Chronic Obstructive Pulmonary Disease
Acronym: ASA-COPD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rolf Ziesche, Professor, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-022123-29
Record Dates: First submitted 2011-03-29; First posted 2011-04-04 (Estimated); Last update posted 2012-12-25 (Estimated); Status verified 2012-12

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ASA (Active Comparator)
  Interventions: Drug: Acetylsalicylic acid
- Placebo (Placebo Comparator)
  Interventions: Drug: Acetylsalicylic acid

INTERVENTIONS:
Drug: Acetylsalicylic acid — 500 mg /day

SUMMARY:
The pathomechanisms of COPD are still not fully understood, and up to now there is no satisfying causal treatment inhibiting the progress of the disease. Available therapy is in most cases symptomatic. Experimental and clinical observations suggest that treatment with ASA might be beneficial in the treatment of COPD in terms of respiratory and lung-functional improvement.

To evaluate the efficacy of ASA as add-on therapy in COPD in comparison to placebo a prospective, randomized, double-blind, placebo controlled study will be conducted. Adult male and female patients (n=74) with proven COPD GOLD grade II-III will be randomized to 2 groups (i.e. 37 patients per group, stratification according to smoking status and gender). They will receive either 500 mg ASA per day or matching placebo over 12 weeks. Primary efficacy endpoints are changes in the lung-functional parameter FEV1 (forced expiratory 1-second volume) after 12 weeks of treatment. Secondary endpoints are the health score of the St. Georges respiratory questionnaire (SGRQ) and Peak-flow (PEF).

ELIGIBILITY:
Inclusion Criteria:

* COPD GOLD II or III

Exclusion Criteria:

* Long term NSAIDS, pregnancy et al.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Change in FEV1 (forced expiratory volume in 1 second) after 12 weeks of treatment | 12 weeks
  lung functional testing

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Ziesche, MD, Professor, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria